CLINICAL TRIAL: NCT04203277
Title: Improving Vaccinations for Young Children (IVY)
Acronym: IVY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth Williams, Assistant Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 190032
Record Dates: First submitted 2019-12-09; First posted 2019-12-18 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Vaccination Refusal
Keywords: vaccine uptake, timely vaccination
MeSH Terms: conditions — Vaccination Refusal

STUDY DESIGN:
Intervention Model Description: Intervention effectiveness on improving vaccination rates will be evaluated using a SW-CRT. 36 Eight practices (clusters) will eventually be randomized to receive the IVY intervention over a 13-month study period. Patients are clustered within practices, and outcomes will be assessed on cross-sectional samples of individuals at each practice at 13 discrete, monthly time points. There will be a baseline block of two months where all practices will be in the control group (Figure 3). Following this, two practices will be randomly assigned to receive the intervention (Group 1). Two months after initiation of IVY in Group 1, two practices will be randomly assigned to receive the intervention in Group 2. This will be continued for 4 total Groups. There will be a five-month block after implementing IVY in all practices where data will continue to be collected after all have been assigned to receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Step Wedge Randomized Group 1 (Experimental): Includes two pediatric practices randomized to the first step of the step-wedge randomized trial
  Interventions: Other: IVY
- Step Wedge Randomized Group 2 (Experimental): Includes two pediatric practices randomized to the second step of the step-wedge randomized trial
  Interventions: Other: IVY
- Step Wedge Randomized Group 3 (Experimental): Includes two pediatric practices randomized to the third step of the step-wedge randomized trial
  Interventions: Other: IVY
- Step Wedge Randomized Group 4 (Experimental): Includes two pediatric practices randomized to the fourth step of the step-wedge randomized trial
  Interventions: Other: IVY

INTERVENTIONS:
Other: IVY — a combination of practice education and quality improvement interventions

SUMMARY:
The IVY project focuses on improving combination 10 vaccine rates for Tennessee children through an educational and quality improvement intervention rolled out through a stepped-wedge cluster randomized trial.

DETAILED DESCRIPTION:
The proposed work seeks to improve Combination 10 vaccination rates for Tennessee children at 2 years of age through the development and implementation of a new program, Improving Vaccination for Young Children (IVY). Through a collaboration with the Cumberland Pediatrics Foundation (CPF), a non-profit company focused on improving health care services for Tennessee's children, investigators plan to adapt and disseminate existing CoVER educational materials for community pediatric providers and clinical staff, and develop and implement targeted quality improvement (QI) initiatives.

A.3. Specific Objectives:

1. Design interactive web-based modules individualized for two groups (pediatric providers and pediatric clinical staff) to educate on key vaccine topics. Modules will include information related to 1) diseases vaccines are targeting, including influenza 2) vaccine contraindications, common misconceptions, and vaccine safety, 3) communication techniques, 4) vaccine schedules and catch up rules, and 5) exemptions, school requirements, and practice dismissal.
2. Design an in-person QI coaching session incorporating key drivers for improved vaccination rates. The session will be developed using the 4Pillars™ Practice Transformation Program (4Pillars™) and will include introduction of 1) acute visits for vaccine catch up, 2) team-based care practices, 3) standing vaccination record review and vaccination orders, and 4) reminder/recall systems.
3. Implement educational modules and QI coaching session at specific time points within the context of a stepped wedge cluster randomized trial (SW-CRT). Combination 10 [(Combo 10)] vaccine rates will be collected monthly from the Electronic Health Record (EHR) of recruited practices for eligible children turning 2 years of age. Vaccine rates will be compared between practices monthly within the SW-CRT design. Rates will also be evaluated by practice over time.

ELIGIBILITY:
Inclusion Criteria:

* pediatric clinics
* serving children at minimum up to age 2
* located in Tennessee

Exclusion Criteria:

-none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Combination 10 vaccination rates in 2 year old children | Assessing change in combination 10 vaccination rates in 2 year old children up to 12 months
  The primary outcome is individual patient-level receipt of all vaccinations [Combo 10 (binary, yes/no)] for children turning 2 years of age in prior month.

SECONDARY OUTCOMES:
Combination 3 vaccination rates in 2 year old children | Assessing change in combination 3 vaccination rates in 2 year old children up to 12 months
  The primary outcome is individual patient-level receipt of all vaccinations [Combo 3 (binary, yes/no)] for children turning 2 years of age
Additional sub analyses of combination 10 vaccination rates (excluding flu vaccine) in 2 year old children | Assessing change in combination 10 vaccination (excluding flu vaccine) rates in 2 year old children up to 12 months
  We will adjust our data and analyze combo 10 vaccination rates minus influenza vaccine.
Additional sub analyses of combination 10 vaccination rates in 2 year old children adjusting for proportion of practice who complete educational training | Assessing how "dose" of educational training affects change in combination 10 vaccination rates in 2 year old children up to 12 months
  We will determine proportion of the practice who completed the educational training and conduct a dose analysis.
Additional sub analyses of combination 10 vaccination rates in 2 year old children adjusting for whether practice represents a community or academic population | Assessing change in combination 10 vaccination rates in 2 year old children up to 12 months, adjusting for educational "dose"
  We will adjust for the bivariate variable of community versus academic population within our analysis model. Community practices are those that are recruited by our partner Cumberland Pediatric Foundation and academic practices are those directly affiliated with Vanderbilt.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Williams, MD, MPH, Principal Investigator — Vanderbilt University
Locations (1):
- Sarah E Williams, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams SE, Adams LE, Sommer EC. Improving Vaccination for Young Children (IVY): A Stepped-Wedge Cluster Randomized Trial. Acad Pediatr. 2021 Sep-Oct;21(7):1151-1160. doi: 10.1016/j.acap.2021.06.001. Epub 2021 Jun 10. PMID 34118498